CLINICAL TRIAL: NCT01252134
Title: The Evaluation of Silicone Hydrogel Lens Wettability With Marketed Lens Care Solutions
Brief Title: Evaluation of Silicone Hydrogel Lens Wettability With Marketed Lens Care Solutions
Acronym: SILVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: RDG10078 / SILVER
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Results first posted 2012-06-11 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-05

CONDITIONS: Contact Lens Wear
Keywords: Soft Contact lens; Multi-purpose solution; Wettability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Synergi, then Biotrue, then OTE (Other): Three lens care systems randomly assigned. Contact lenses were pre-soaked overnight prior to insertion, then worn for 8 hours, with a minimum two-day washout between each wear period.
  Interventions: Device: Biotrue multipurpose solution; Device: Sauflon Synergi multipurpose solution; Device: OTE Elements multipurpose solution; Device: Silicone hydrogel contact lenses (Acuvue Advance)
- Synergi, then OTE, then Biotrue (Other): Three lens care systems randomly assigned. Contact lenses were pre-soaked overnight prior to insertion, then worn for 8 hours, with a minimum two-day washout between each wear period.
  Interventions: Device: Biotrue multipurpose solution; Device: Sauflon Synergi multipurpose solution; Device: OTE Elements multipurpose solution; Device: Silicone hydrogel contact lenses (Acuvue Advance)
- Biotrue, then OTE, then Synergi (Other): Three lens care systems randomly assigned. Contact lenses were pre-soaked overnight prior to insertion, then worn for 8 hours, with a minimum two-day washout between each wear period.
  Interventions: Device: Biotrue multipurpose solution; Device: Sauflon Synergi multipurpose solution; Device: OTE Elements multipurpose solution; Device: Silicone hydrogel contact lenses (Acuvue Advance)
- Biotrue, then Synergi, then OTE (Other): Three lens care systems randomly assigned. Contact lenses were pre-soaked overnight prior to insertion, then worn for 8 hours, with a minimum two-day washout between each wear period.
  Interventions: Device: Biotrue multipurpose solution; Device: Sauflon Synergi multipurpose solution; Device: OTE Elements multipurpose solution; Device: Silicone hydrogel contact lenses (Acuvue Advance)
- OTE, then Biotrue, then Synergi (Other): Three lens care systems randomly assigned. Contact lenses were pre-soaked overnight prior to insertion, then worn for 8 hours, with a minimum two-day washout between each wear period.
  Interventions: Device: Biotrue multipurpose solution; Device: Sauflon Synergi multipurpose solution; Device: OTE Elements multipurpose solution; Device: Silicone hydrogel contact lenses (Acuvue Advance)
- OTE, then Synergi, then Biotrue (Other): Three lens care systems randomly assigned. Contact lenses were pre-soaked overnight prior to insertion, then worn for 8 hours, with a minimum two-day washout between each wear period.
  Interventions: Device: Biotrue multipurpose solution; Device: Sauflon Synergi multipurpose solution; Device: OTE Elements multipurpose solution; Device: Silicone hydrogel contact lenses (Acuvue Advance)

INTERVENTIONS:
Device: Biotrue multipurpose solution — Contact lens care solution
Device: Sauflon Synergi multipurpose solution — Contact lens care solution
Device: OTE Elements multipurpose solution — Contact lens care solution
Device: Silicone hydrogel contact lenses (Acuvue Advance) — Commercially marketed contact lenses
  Other Names: Acuvue® Advance™

SUMMARY:
The purpose of this study is to assess ex vivo wettability of a commonly prescribed silicone hydrogel (SiH) contact lens with three marketed contact lens care solutions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Soft contact lens wear on a daily wear basis
* Able to wear lenses at least 8 hours
* Generally healthy with normal ocular health
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Use of additional lens cleaners
* Known sensitivities to any ingredient in any of the study products
* History of ocular surgery/trauma within the last 6 months
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled from one Canadian study center.
Period: Period 1, 8 Hours
Arm/Group | Synergi, Then Biotrue, Then OTE | Synergi, Then OTE, Then Biotrue | Biotrue, Then OTE, Then Synergi | Biotrue, Then Synergi, Then OTE | OTE, Then Biotrue, Then Synergi | OTE, Then Synergi, Then Biotrue
Started | 3 | 4 | 3 | 5 | 3 | 4
Completed | 3 | 3 | 2 | 5 | 3 | 4
Not Completed | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Personal Reasons | 0 | 1 | 1 | 0 | 0 | 0
Period: Period 2, 8 Hours
Arm/Group | Synergi, Then Biotrue, Then OTE | Synergi, Then OTE, Then Biotrue | Biotrue, Then OTE, Then Synergi | Biotrue, Then Synergi, Then OTE | OTE, Then Biotrue, Then Synergi | OTE, Then Synergi, Then Biotrue
Started | 3 | 3 | 2 | 5 | 3 | 4
Completed | 3 | 3 | 2 | 5 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3, 8 Hours
Arm/Group | Synergi, Then Biotrue, Then OTE | Synergi, Then OTE, Then Biotrue | Biotrue, Then OTE, Then Synergi | Biotrue, Then Synergi, Then OTE | OTE, Then Biotrue, Then Synergi | OTE, Then Synergi, Then Biotrue
Started | 3 | 3 | 2 | 5 | 3 | 4
Completed | 3 | 3 | 2 | 5 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: All enrolled participants
Arm/Group | Overall
Number analyzed (Participants) | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 24.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Ex Vivo Contact Angle
Description: Study lens was removed from the eye according to protocol-specified procedures. The OCA15 Dynamic Contact Angle Instrument was used to observe, record, and calculate contact angle measurements. The measurements from the right eye and left eye were averaged. A lower contact angle measurement indicates a more wettable lens.
Time Frame: 8 hours
Population: This reporting group includes all participants who completed the study, minus one response in Synergi group due to a measurement error.
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Synergi; Bio-True; OTE Elements: Contact lenses were pre-soaked overnight prior to insertion, then worn for 8 hours.
Arm/Group | Synergi | Bio-True | OTE Elements
Number analyzed (Participants) | 19 | 20 | 20
degrees | 104.8 (2.4) | 104.9 (3.7) | 103.3 (5.4)

2. Secondary Outcome: Subjective Comfort
Description: Subjective comfort was assessed by the participant on a scale of 0 to 100, with 0 being very poor comfort and 100 being excellent comfort. The ratings for the right eye and left eye were averaged.
Time Frame: 8 hours
Population: This reporting group includes all participants who completed the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Synergi | Bio-True | OTE Elements
Number analyzed (Participants) | 20 | 20 | 20
Units on a scale | 87.3 (7.9) | 87.3 (10.2) | 86.4 (15.0)

3. Secondary Outcome: Corneal Staining Type
Description: Five regions of the cornea (central, inferior, temporal, superior, and nasal) were evaluated for staining using cobalt light and a #12 Wratten filter. The type of staining was recorded on a scale of 0 to 100 for each corneal region with 0-none, 25=micropunctate, 50=macropunctate, 75=coalescent, and 100=patch. The five regions for each eye were averaged, and the eyes were averaged.
Time Frame: 8 hours
Population: This reporting group includes all participants who completed the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Synergi | Bio-True | OTE Elements
Number analyzed (Participants) | 20 | 20 | 20
Units on a scale | 5.4 (8.4) | 8.8 (8.4) | 3.0 (4.7)

4. Secondary Outcome: Corneal Staining Extent
Description: Area (extent) of corneal staining was estimated for each of the five regions of the cornea as a percentage i.e., 0%=no staining in the region and 100%=staining covering the entire region). A staining area percentage was calculated for each eye based on the average staining area measured across all five regions, and the eyes were averaged.
Time Frame: 8 hours
Population: This reporting group includes all participants who completed the study.
Measure: Mean (Standard Deviation); unit: percentage of cornea
Arm/Group | Synergi | Bio-True | OTE Elements
Number analyzed (Participants) | 20 | 20 | 20
percentage of cornea | 0.7 (0.8) | 3.1 (3.8) | 0.9 (4.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the trial: 24-NOV-2010 to 8-FEB-2011.
Description: This reporting group includes all enrolled and exposed participants
Arm/Group | Synergi | Bio-True | OTE Elements
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other